CLINICAL TRIAL: NCT04661059
Title: Study of Late-foetal Human Organ Development
Status: Recruiting | Type: Observational
Sponsor: University College London Hospitals (Other)
Responsible Party: Principal Investigator, Marko Nikolic, Principal Investigator, University College London Hospitals
Other Study IDs: 253088
Record Dates: First submitted 2020-12-01; First posted 2020-12-09 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Congenital Disorders
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Knowledge about abnormal organ development is important to understand pathology and to develop novel treatment approaches for individuals with congenital and acquired disease. Most of our current understanding is based on examination of tissues from the embryo and early fetus, collected from women undergoing termination of pregnancy in the first trimester (third) of pregnancy. There is very little known about normal and abnormal organ development from a developmental perspective during the crucial last two-thirds of pregnancy when much remodelling of fetal tissues occurs. We aim to collect tissue from a variety of developing fetal organs in the last two-thirds of pregnancy from women who decide to undergo a termination of pregnancy and who wish to undergo a clinical fetal postmortem (PM) examination.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old pregnant women who attend the Fetal Medicine Unit for concerns about a fetal abnormality where they decide to proceed to termination of pregnancy

Exclusion Criteria:

* Screening labs positive for maternal HIV, Hepatitis B and Hepatitis C, Chlamydia and Herpes.
* Subject unable to make an informed decision about termination of pregnancy.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: As above
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-02-03 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2040-12-31 (Estimated)

PRIMARY OUTCOMES:
Cellular maturity | Immediately after tissue collection
  Immunofluorescence staining

CONTACTS AND LOCATIONS:
Locations (1):
- University College Hospitals NHS Foundation Trust, London, United Kingdom